CLINICAL TRIAL: NCT02314039
Title: Psychological Factors in Acne: A Focus on Psychological Trauma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Edinburgh Napier University (Other)
Responsible Party: Principal Investigator, Dr Zoe Chouliara, Dr Zoe Chouliara, Edinburgh Napier University
Other Study IDs: 14-SS-1072
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This cross sectional questionnaire based study will aim at exploring psychological factors at play in the experience of acne, and their association with perceived and clinical severity. We will focus in particular on the role of psychological trauma in the patients with acne and their wellness. This project is being undertaken as part of a wider developing initiative in the Dermatology Department within NHS Tayside, which aims at identifying and consequently addressing the psychological needs of their patients. Participants will be consecutive patients with acne aged at least 18 years old, seen in the outpatient clinics of the Dermatology Department in NHS Tayside. Potential participants will be informed about the research by their clinician during an outpatients appointment and if interested, given an information sheet and consent form to review. Verbal consent will be sought by the clinician to give the potential participant's contact details to the Chief Investigator (CI)/Research Assistant (RA). If agreeable, the CI/RA will contact the potential participant after at least 24 hours to arrange a mutually agreed time for meeting. If the potential participant are still keen to participate and has read the information sheet, fit our inclusion criteria, are not deemed to be distressed by their attending clinician and want to take part, they will be included. Participants will complete a number of standardised questionnaires and a demographics information sheet in the outpatients' clinic with the CI/RA present. The questionnaires include questions on psychological trauma history and symptomatology, general psychological distress, appearance related distress and perceived severity of condition. Clinical severity of their acne will be obtained from patient files after questionnaire completion by NHS staff. Participants will also be given a debrief letter and additional forms of support and information to take home with them. Participants will not be contacted for follow-up.

DETAILED DESCRIPTION:
The research questions are as follows:

1. What is the association between psychological trauma symptoms, and perceived/clinical severity of the condition?
2. What are the levels of psychological trauma symptoms exhibited in patients with acne?
3. What are the associations between traumatic history (in childhood and adulthood), current traumatic symptoms exhibited and perceived/clinical severity?
4. What is the association between psychological trauma symptomatology, trauma history, general psychological distress, appearance-related distress and perceived/clinical severity?

Design: A quantitative cross--sectional design will be used. Five self-report, standardised questionnaires will be completed by participants and assisted by the Chief Investigator (CI) or the Research Assistant (RA) to the study. The questionnaires contains measures on:

psychological trauma history; perceived severity of acne; general appearance--related distress; and depression, stress and anxiety.

Basic demographics will be collected by asking participants to also complete a Demographics Information sheet (measuring age, gender, time since diagnosis etc.). Information on objective severity of acne will be provided by staff (e.g. named specialist nurse of consultant dermatologist for each clinical site). Information on objective severity is routinely measured in dermatology clinical practice and such information will be available in file for each patient.

Participants: The population sample will be recruited from NHS Tayside dermatology departments, i.e. Ninewells, Strathcathro and Perth Hospital.

Procedure & recruitment: The CI will liaise with Principal Investigator (PI), Dr Andrew Affleck, and arrange to present the study to clinical staff teams in each of the names clinical sites. The CI and RA will meet with relevant staff at the recruitment sites to discuss the purpose and nature of the study prior to and throughout the recruitment and data collection process. The researchers will also commit to present the findings of the research to the participating clinical teams when the study is completed.

Pre-Testing Phase: Information packs regarding the study will be provided to clinical staff at the recruitment sites. The information packs will include: background information and purpose of the study, and participant exclusion/inclusion criteria. Staff at the recruitment sites will be asked to identify suitable participants who meet the criteria outlines in the study. The CI and RA will not be required to review patient records.

Suitable participants will be initially approached by a familiar member of staff. The clinician will inform the potential participant about the research, introduce the study with an explanation of what would be involved in taking part and the potential participants will be asked if they would be interested in considering participation in the study. If interest is expressed, the potential participants will be provided with further information, including a Participant Information Letter and a consent form. The potential participant will be given the opportunity to ask the clinician questions about the study. Verbal consent will be obtained from the potential participant to pass their details onto the CI/RA so a meeting can be arranged. Contact details will be given to the CI/RA either in person or via telephone.

The potential participant will be given at least 24 hours to further consider the study before the CI/RAcalls to arrange a meeting. A meeting will be arranged, at a mutually agreed time at the clinic to meet each potential participant. The meeting will be arranged either at the time of their follow up appointment or at another agreed time which is convenient for the potential participant. The time between arranging the meeting and the actual meeting provides the potential participants with additional time to consider participation in the study. On the day of the scheduled appointment, the CI/RA will liaise with clinical staff in charge of the care of the patient to check if the participant still meets eligibility criteria and if they still wish to meet with the CI/RA. The CI/RA to the study will meet with the potential participant to verbally review the Participant Information Letter and provide an opportunity for the participants to ask any questions about the study. This will help ensure that the potential participant understands the information presented and are able to provide informed consent. If the potential participant would like to further consider participation, a further meeting will be arranged. If the CI/RA contacts clinical staff and is informed that it is not appropriate to meet with the participant at this time, for example, if the potential participant is distressed or unwell on the day, the meeting will not take place that day. However, if the participant still meets the eligibility criteria at a later date and wishes to take part, the appointment can be rescheduled.

Testing Phase: Further to reviewing the Patient Information Letter, if the participant meets the inclusion criteria and provides agreement to take part, a signed informed consent will be obtained. After the CI/RA has obtained signed consent from the participant, the study measures will be completed. The CI/RA will remain present throughout the testing phase to provide appropriate assistance with the completion of the measures. The CI/RA will offer to read the questions and record the participant's responses in case the participant has literacy difficulties or visual difficulties. The participant will also have a copy of the questionnaires to view when they are being completed. Participants will be offered breaks, however, if they become fatigued, they will also be offered to continue the testing on another date or withdraw from the study. If for any other reason the participant becomes distressed or the CI/RA deems the participant as unable to understand the study related information or questionnaires, the testing will be discontinued and appropriate action in line with clinical practice will be taken.

Post-Testing Phase: Following the completion of the testing phase, each participant will be given the opportunity to discuss their participation in the study and raise concerns of difficulties they experienced during completion of the study. Participants will also be made aware that they can discuss their experience with a named independent person, whose contact will be clearly mentioned in the Debrief. Should participants become distressed or highlight concerns, the CI will use her clinical skills, as a Practitioner Counselling and Health Psychologist and Psychotherapist Counsellor. The RA to the study will be supervised closely and frequently by the CI. The RA is knowledgeable in the area of skin disorders and acne in particular at Masters level, and has worked in many clinical studies before as part of her post with the Mental Health Research Network. She also has a certificate in Good Clinical Practice (June, 2014). When data collection is carried out by the RA, the RA will perform her duty of care at all times and will follow good practice and ethics for research guidelines. Any concerns the RA has, she will discuss with the CI immediately, who will be available to be contacted during meeting with participants and will provide her with further guidance about which course of action should it be necessary. If distress escalates and the CI is unavailable, the RA will contact appropriate clinical staff (e.g. Dr Andrew Affleck, a named nurse or another consultant dermatologist on site) for advice and input, if necessary. Potential participants will be made aware of these stages and limitations to confidentiality prior to consenting to take part. A Patient Information Sheet will be completed by the patient along with the rest of the measures.

Clinical severity score will be obtained from patient files by clinical staff. The CI and the RA will have no contact with patient files. The study packs will be anonymised prior to administration, i.e. a participant code will be printed on every page of the pack, including the participant information letter, consent form and participant debrief. Consent forms will be separately handed to Dr Andrew Affleck in person and will be securely kept locked in a cabinet on NHS Tayside premises. Completed questionnaires will be separated from consent forms immediately after completion and questionnaires will be kept separately on Edinburgh Napier University premises. From that point on, the CI and the RA will have no access to the consent forms. Only Dr Affleck will have access to the consent forms. Anonymised data will be entered on a electronic statistical package (SPSSX) that will be password protected. As part of the governance of the study, we have now put in place, Professor Kevin Power, Head of Psychological Services, NHS Tayside, has agreed to monitor the clinical governance of this research study. The researchers, i.e. CI and the RA, will score the psychological trauma screening questionnaires on the spot. If the participants are identified in the testing phase as scoring within the clinical range in post-traumatic symptoms, the CI will notify the consultant dermatologist in charge of this patient, who will then notify Prof. Power. Prof. Power will ensure that such patients enter an appropriate clinical pathway via appropriate referral. Participants will be notified of this governance as part of their information letter and participant debrief.

Measures: The measures will be administered by the CI or the RA by paper and pencil or verbally, if required.

ELIGIBILITY:
Inclusion Criteria:

* Patients in NHS Tayside in one of the three participating dermatology outpatient departments
* Aged 18 years old or older
* Attending the clinic for acne
* Fluent in speaking and understanding English
* Deemed by qualified clinical staff as routine practice, as able to give informed consent form

Exclusion Criteria:

* Individuals who have a learning disability or organic disorder that would impair their ability to provide informed consent or understand and respond to the questionnaires
* Under the influence of illicit substances at the time of administration of the questionnaires
* In a distressing state, as judged by clinical staff and/or the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population sample will be recruited from NHS Tayside dermatology departments, i.e. Ninewells, Stracathro, and Perth Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Psychological trauma symptoms | This outcome will be measured once during the 6 month recruitment period. All outcomes will be measured at the same timepoint. This timepoint is expected to last no longer than 2 hours.
  This will be measured using the ICD 11 Trauma Questionnaire (Knefel & Lueger-Schuster, 2013) and will be used to answer all the research questions

SECONDARY OUTCOMES:
Perceived severity of acne | This outcome will be measured once during the 6 month recruitment period. All outcomes will be measured at the same timepoint. This timepoint is expected to last no longer than 2 hours.
  This will be measured by the Cardiff Acne Disability Index (Motley & Finlay, 1992) and will be used to answer research questions 1, 3 and 4.
Clinical severity of acne | This outcome will be measured once during the 6 month recruitment period. All outcomes will be measured at the same timepoint. This timepoint is expected to last no longer than 2 hours.
  This is measured as a part of routine assessment in all acne patients attending dermatology departments. The information can be found in patients' files and is recorded in the format 'mild, moderate or severe acne'. This information will be used to answered research questions 1, 3 and 4.
Childhood traumatic history | This outcome will be measured once during the 6 month recruitment period. All outcomes will be measured at the same timepoint. This timepoint is expected to last no longer than 2 hours.
  This will be measured using the Childhood Trauma Questionnaire (Bernstein et al., 1994) and will be used to answer research questions 3 and 4.
Adult traumatic history | This outcome will be measured once during the 6 month recruitment period. All outcomes will be measured at the same timepoint. This timepoint is expected to last no longer than 2 hours.
  This will be measured using Life Events Checklist (Blake et al, 1995) and will be used to answer research questions 3 and 4.
General psychological distress | This outcome will be measured once during the 6 month recruitment period. All outcomes will be measured at the same timepoint. This timepoint is expected to last no longer than 2 hours.
  This will be measured using the DASS 21(Lovibond & Lovibond, 1995) and will be used to answer research question 4.
Appearance-related distress | This outcome will be measured once during the 6 month recruitment period. All outcomes will be measured at the same timepoint. This timepoint is expected to last no longer than 2 hours.
  This will be measured using the Derriford Appearance Scale (DAS) (Carr et al., 2000) and will be used to answer research question 4.

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Chouliara, PhD, Principal Investigator — Edinburgh Napier University